CLINICAL TRIAL: NCT06069102
Title: OPT-BP: Optimal Blood Pressure Treatment Thresholds Following a Hypertensive Disorder of Pregnancy: A Pilot Trial
Brief Title: Optimal Blood Pressure Treatment Thresholds Postpartum
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alisse Hauspurg (Other)
Responsible Party: Sponsor-Investigator, Alisse Hauspurg, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY23060147
Record Dates: First submitted 2023-09-28; First posted 2023-10-05 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-06

CONDITIONS: Hypertensive Disorder of Pregnancy; Pre-Eclampsia; Hypertension; Eclampsia; Gestational Hypertension; Cardiovascular Diseases; Toxemia; Pregnancy Complications; Vascular Diseases; Hypertension, Pregnancy Induced; Hypertension;Pre-Eclamptic
Keywords: Hypertension
MeSH Terms: conditions — Toxemia; Pre-Eclampsia; Hypertension; Eclampsia; Hypertension, Pregnancy-Induced; Cardiovascular Diseases; Pregnancy Complications; Vascular Diseases

STUDY DESIGN:
Intervention Model Description: The investigators will conduct a prospective single site, single-blinded, parallel randomized control trial in which individuals diagnosed with HDP will be randomized to usual care or tight blood pressure control for therapeutic intent. Subjects will undergo 3 study visits (1 in-person and 2 remote) involving BP measurements, blood draws, and/or questionnaires.
Who Masked: Outcomes Assessor
Masking Description: Once randomization is complete, there will be no blinding of participants, care providers or investigators. Outcomes assessors will be masked to intervention arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Usual Care Group (Active Comparator): Standard of care BP medication will usually be started if a subject's BP consistently exceeds 150/100 mmHg at any point.
  Interventions: Drug: Usual care
- Intervention (Tight Blood Pressure Control) Group (Experimental): BP medication will be started if a subject's hospital BP consistently exceeds 140/90 mmHg or her home BP consistently exceeds 135/85 mmHg.
  Interventions: Drug: Tight blood pressure control

INTERVENTIONS:
Drug: Usual care — The usual care group will be given anti-hypertensive medications (i.e. beta blocker, calcium channel blocker, etc) if a subject's BP consistently exceeds 150/100 mmHg consistently.
  Arms: Usual Care Group
Drug: Tight blood pressure control — The intervention group will be initiated on blood pressure medications (i.e. beta blocker, calcium channel blocker, etc) if a subject's hospital BP consistently exceeds 140/90 mmHg or home BP consistently exceeds 135/85 mmHg.
  Other Names: Tight control
  Arms: Intervention (Tight Blood Pressure Control) Group

SUMMARY:
The objective of this research project is to conduct a single-site pilot trial within our institution's clinical remote blood pressures (BP) management program to assess the feasibility and effect of tight blood pressure control versus usual care in the immediate postpartum period after a hypertensive disorder of pregnancy (HDP).

The investigators' central hypothesis is that tight blood pressure control will be feasible and acceptable to postpartum individuals and will result in lower BP at six months postpartum and a reduction in postpartum hospital readmissions. Subjects will undergo 3 study visits (1 in-person and 2 remote) involving BP measurements, blood draws, and/or questionnaires. Up to 60 adult subjects will be enrolled at Magee-Women's Hospital.

DETAILED DESCRIPTION:
The investigators will determine the feasibility of conducting a randomized controlled trial of tight blood pressure control (<135/85 mmHg on home BP monitoring) vs. standard of care (<150/100 mmHg on home BP monitoring) in postpartum individuals following a HDP with assessment of individuals who are eligible, enrolled, and remain in the study until six weeks postpartum. Individuals who are retained in the study for 6 months postpartum. Lastly, investigators will analyze effect outcomes to inform the sample size for a subsequent large-scale randomized trial. This will be done through analysis of mean arterial pressure (MAP), systolic blood pressure, and diastolic blood pressure of participants at 6 weeks and at 6 months postpartum. The study will be conducted on the postpartum unit of Magee-Womens Hospital. Participants will be enrolled at the time of postpartum hospitalization with study visit #1 occurring in the hospital. At this study visit, participants will be administered questionnaires, will provide a blood sample, and BP will be measured. Study visit #2 will be a remote study visit conducted via telemedicine or a telephone call at 6 weeks postpartum. At this visit, participants will provide questionnaires and blood pressure data. Study visit #3 will be a remote study visit conducted via telemedicine or a telephone call at 6 months postpartum. At this visit, participants will again provide questionnaires and blood pressure data.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum individuals ≥18 years old
* Preeclampsia or gestational hypertension diagnosis (complying ACOG criteria)
* Enrolled in remote BP management program.

Exclusion Criteria:

* Pre-pregnancy hypertension
* Pre-pregnancy diabetes
* Maternal cardiac disease
* Chronic kidney disease

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Percent of participants eligible, enrolled and retained (feasibility) | Baseline to approximately 6 months postpartum
  To determine if a randomized controlled trial of tight blood pressure control (<135/85 mmHg on home blood pressure monitoring) vs. standard of care (<150/100 mmHg on home blood pressure monitoring) in postpartum individuals following a hypertensive disorder of pregnancy (HDP) is feasible.

SECONDARY OUTCOMES:
Anti-hypertensive medication use (efficacy) | 6 months postpartum
  Anti-hypertensive medication use
Anti-hypertensive medication use | 6 weeks postpartum
  Anti-hypertensive medication use
Mean arterial pressure (efficacy) | 6 months postpartum
  Mean arterial pressure (systolic BP + 2*diastolic BP / 3)
Mean arterial pressure | 6 weeks postpartum
  Mean arterial pressure (systolic BP + 2*diastolic BP / 3)
Systolic blood pressure | 6 months postpartum
  Mean systolic blood pressure
Diastolic blood pressure | 6 months postpartum
  Mean diastolic blood pressure
Diastolic blood pressure | 6 weeks postpartum
  Mean diastolic blood pressure
Change in MAP | Enrollment to 6 weeks postpartum
  Change in mean arterial pressure (systolic BP + 2*diastolic BP / 3)
Change in systolic BP | Enrollment to 6 weeks postpartum
  Change in systolic BP
Change in diastolic BP | Enrollment to 6 weeks postpartum
  Change in diastolic BP
Proportion of participants with readmissions | Enrollment through six months postpartum
  Postpartum hospital readmissions
Proportion of participants with ER visits | Enrollment through six months postpartum
  Emergency room visits

CONTACTS AND LOCATIONS:
Overall Officials: Alisse K Hauspurg, MD, Principal Investigator — UPMC Magee Women's Hospital
Locations (1):
- University of Pittsburgh Magee-Womens Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data (including data dictionaries) will be shared at the direction of the primary investigator. Data will include blood pressure, weight, demographics, physical activity, and pregnancy related information. Additional documents (such as the study protocol) will be made available. The dataset for our project will be prepared according to requirements for and stored on the Clinicaltrials.gov data repository. Per the NIH guidelines, the dataset will be submitted to the program officer within a year after the outcomes are published and no later than 3 years after the end of clinical activities.
Supporting Information: Study Protocol
Time Frame: Within a year after outcomes are published and no later than 3 years after the end of clinical activities.
Access Criteria: NHLBI data repository request process
URL: https://biolincc.nhlbi.nih.gov/home/